CLINICAL TRIAL: NCT05785455
Title: Efficacy Of Pain Neuroscience Communication, Motivational Interviewing And Cognitive Exercise Therapy In Patients With Chronic Neck Pain
Brief Title: Pain Education, Motivational Interviewing and Exercise in Chronic Neck Pain
Acronym: COGMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI21/01261
Record Dates: First submitted 2022-11-15; First posted 2023-03-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Neck Pain
Keywords: Chronic pain; Pain neuroscience education; Exercise therapy; Neck pain; Motivational interviewing
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Subjects will receive a health education program during 5 group sessions of 60 minutes, taught by physical therapists without training in pain neuroscience education.
  All patients will receive 5 sessions, regardless of the group they belong to. Group education sessions will be in groups (of 5-6 patients), respecting the safety distance. Group sessions will be held in person, in small groups, at the health center, on a weekly basis. Both groups will receive online monitoring of the exercise program. An image with more information about the intervention and control is attached in Annex 2.
  Interventions: Other: Usual Care
- COGMO Intervention (Experimental): Each subject will receive. a first individual session to assess their beliefs about pain and coping strategies, combining motivational interviewing and pain neuroscience education techniques, followed by 4 group sessions of 60 minutes, focused on the neurophysiology of pain and self-efficacy techniques in pain control, emphasizing . in two-way communication and followed by cognition targeted exercise therapy. These sessions will be taught by physiotherapists with specific training in motivational interviewing, pain neuroscience education and cognition targeted exercise
  Interventions: Other: COGMO Intervention

INTERVENTIONS:
Other: COGMO Intervention — Group sessions in which each patient, after motivational interviewing sessions will follow a goup education in pain neuroscince program followed by a cognition targeted exercise therapy
  Arms: COGMO Intervention
Other: Usual Care — Usual Primary Care health education and treatment for patients with chronic neck pain
  Arms: Usual care

SUMMARY:
Objectives: To evaluate the effectiveness of a complex intervention (COGMO intervention) compared with routine clinical practice in primary care physiotherapy to improve the intensity, severity of pain, and cervical disability in patients with chronic neck pain.

Methodology: Design: Pragmatic cluster randomized trial with 12-month follow-up. The unit of randomization is the physiotherapist and the unit of analysis the patient.

Scope: Madrid Primary Care health centers. Subjects: Patients 18-65 years old, with neck pain (> 3 months), moderate-severe (>30 mm in visual pain scale). Sample size: 142 patients (71 per branch).

Sampling: consecutive of patients who are referred from the family doctor to the Primary Care physiotherapist. Intervention: COGMO Intervention Group (3 components: pain neuroscience communication, motivational interviewing and cognition targeted exercise therapy). Control group: Health education program. Variables: Main: Decrease in intensity of pain: yes / no (> = 30mm on the visual pain scale). Secondary: Related to pain (severity of pain, modulation conditioned to pain, temporal summation, decrease in the disability index, related to psycho-emotional-social aspects: decrease in fear / avoidance behaviour, decrease in kinesiophobia (TSK) and Catastrophism (PCS). Quality of life (Euroqol). Sociodemographic, other treatments, adherence to intervention. Data collection: Baseline visit and 3 follow-up visits (3,6,12 months).

Statistical analysis: Intention-to-treat analysis. Difference in the percentage of subjects who achieve success in the main variable at 12 months in the COGMO group compared to control group. A GEE logit model to adjust for other factors.

DETAILED DESCRIPTION:
Data management

Typology, format and ownership of data: The data to be collected are individual patient variables that will be collected after inclusion in the study and signing of the informed consent. The variables have been detailed in the methodology section and in Annex 1 (questionnaires). The information will be collected through a clinical interview and complementary examination tests.

Repository and data access procedures. Security: The information collected will be incorporated by the researchers into an electronic data collection notebook (CRDe), which will assign a unique code to each patient, and in which there will be no reference to the identity of the subjects. Each researcher will keep the list of their included patients, with the link between code and affiliation on a secure site. Access to the CRDe will be done with a user ID and password, and it will be hosted on the research/innovation server of the Primary Care Assistance Management/ Primary Care Biosanitary Research and Innovation Foundation (FIIBAP) in Madrid. The results will be disseminated in scientific forums, congresses, scientific publications and in social media, maintaining the confidentiality and rights of the participants. In no case will data that allows them to be identified be published. In order to maximize access and reuse of scientific data generated by the project, the results and the anonymized database will be published openly, always within the framework of legal regulations.

Ethical and legal aspects: The trial will respect the basic ethical principles of autonomy, beneficence, justice and non-maleficence and will follow the standards of Good Clinical Practice and the principles set forth in the latest declaration of Helsinki and the Oviedo Convention (1997). ). Study subjects will be fully informed of the study, and will only be included if they provide written informed consent, clearly detailing post-hoc data use. With regard to the treatment, communication and transfer of data, it will be done in accordance with the provisions of the RGPD (EU Regulation) 2016/679 of the European Parliament and of the Council, of April 27, 2016 and the LOPDGDD 3/2018, of December 5th.

Hypothesis

Conceptual hypothesis: In patients with chronic neck pain, a complex multicomponent intervention (based on pain neuroscience education, motivational interviewing and cognitive exercise therapy: "COGMO intervention") performed by primary care physical therapists will increase. the proportion of patients with clinical improvement in pain intensity, compared with a standard exercise health education programme.

Operative hypothesis: In patients with chronic neck pain, a complex "COGMO" intervention will achieve an absolute difference in the percentage of patients who achieve a clinical improvement in pain intensity (at least 30mm in the long-term VAS: 12 months), which will be at least 25% more, in the intervention group compared to the group control.

Objectives

Main goal

Evaluate the effectiveness of a complex intervention "COGMO Intervention" based on education in neuroscience of pain, motivational interviewing and cognitive exercise therapy compared with practice routine clinical practice in physiotherapy (health education with exercises), to improve the intensity of pain, in patients wit Chronic Neck Pain at 12 months of follow-up.

Secondary Objectives

To evaluate the effectiveness of the COGMO intervention against usual therapy with health education at 3, 6 and 12 months to improve: o Pain: intensity, severity, total and distal mechanical hyperalgesia, pain conditioned modulation, changes in pain-free joint range of motion (ROM) and motor control. o Psychosocial aspects: depressive symptoms, anxiety, kinesophobia, catastrophism, fear of pain. o Patient-reported outcomes (PROMS): health-related quality of life. To describe the adherence to the COGMO intervention and the degree of satisfaction of the patients with the therapy received in both groups.

Methodology

Design: Pragmatic randomized cluster clinical trial with 12-month follow-up. The unit of randomization is the physiotherapy professional and the unit of analysis is the patient.

Population: Patients with chronic neck pain under follow-up in Primary Care Centers (PCC).

Scope: 14 PCC of the Community of Madrid (Arroyo de la Vega, Valdelasfuentes, Colmenar Viejo Sur, Dr. Castroviejo, Ciudades, Isabel II, Barrio del Pilar, Colmenar de Oreja, La Cabrera, Mirasierra, Ibiza, Miraflores, Espronceda and Los Yébenes.

Sample size: According to two systematic reviews, chronic neck pain with manual physiotherapy treatment improves by 11% compared to 29% in the control group. Expecting to find a difference in percentages of patients who achieve a clinically significant decrease in pain (at least 30 mm on the visual scale), of 25% more patients in the COGMO intervention group than in the control group, for a level of confidence 95% and 80% power, 58 subjects would be needed in each group. Considering that the average size of the cluster of patients per physiotherapist is 6 patients, and for an intercalate correlation coefficient of 0.02, the design effect will be. of 1.1 [(DE=1+(6-1)*0.02=1.1, (58+58)*DE(1.1)] the necessary sample size would be 128 patients, overestimating due to possible losses of 10%, the final size is 142 patients (71 per branch).

Sampling: consecutive of the patients included in the waiting list of patients referred to the Unit of Physiotherapy in each health center.

Recruitment: Of professionals: the research team already has an associated clinical group of at least 29 physiotherapists. Patients: They will be selected from the list of patients (provided by the health service) who meet the inclusion criteria for each professional's quota. Subsequently, each physiotherapist offer. Consecutively, the participation of patients from the received list, until completing a number of 5-6 per physiotherapist. When the patient agrees to participate, the physiotherapist will inform. in detail about the study, confirm. inclusion/exclusion criteria and patient acceptance with the signing of the informed consent. If the patient does not accept, data on age, sex and reason for refusal will be collected.

The patient recruitment period is estimated at one year and the follow-up of each patient lasts 12 months. from the end of the COGMO or EPS intervention.

Randomization: The randomization unit is the physical therapists who will participate in the study and the analysis are the patients. It will be done. using the module for assigning subjects to treatment of the program Epidat 4.1, considering as treatment the intervention to study COGMO and as control the project of EPS exercises. To obtain the same number of professionals in each group (intervention and control) it will be used. the option of balanced groups. Once the physiotherapist has been assigned to a study group, all patients recruited by him/her will be included in that group. The assignment will be. carried out centrally by the Research Support Unit of the AP Madrid Healthcare Management. It will be done. after each physiotherapist has included and made the selection of patients and the external evaluators have collected the variables of the baseline visit. Subsequently, each MF will receive. the information of the study group to which it has been assigned.

Physiotherapists assigned to the intervention group will receive training in the intervention and those in the control group will access the project. At the end of the trial, interested physiotherapists in the control group will be able to receive training in the COGMO intervention.

Blinding: Due to the characteristics of the study, it is not possible to blind patients or physiotherapists. who will deliver the COGMO intervention or control. The assessors of the outcome variables will be blinded. In addition, at the end of each evaluation they will be examined. the success of blinding the assessor by asking him to indicate the participant group assignment, including percent certainty (50% certainty equals pure guess).

The people in charge of the analysis of results will be blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosed with chronic neck pain, according to the death of the IASP (International Association for the Study of Pain) with duration of pain greater than 3 months and referred to Physiotherapy by their Family doctor.
* Score on the Neck Disability Index (IDC) questionnaire equal to or greater than 20% (10/50).
* Pain intensity at the moment in the cervical region equal to or greater than 30mm on the visual analog scale.

  * Sign informed consent

Exclusion Criteria:

* Neuropathies and/or radiculopathies, other pathologies or comorbidities that may contraindicate the therapies to be applied, severe depression, rheumatic, inflammatory diseases, cancer, suspected fibromyalgia, systemic diseases, serious psychological disorders, neck pain secondary to an accident of traffic.
* Criteria for referral to surgery or failed spinal surgery.
* Inability to read, understand and complete questionnaires; o understand and follow verbal commands.
* Have received physical therapy in the last 3 months.
* Have any pending legal action (for example: compensation for injury).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-14 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The visual analog scale (VAS). This is a 100-mm line with "no pain" on the left side of the line and "worst pain imaginable" on the right side. The patient marks the intensity of her pain on a flat line, which allows observing the result obtained on the 100 mm line, being able to quantify her pain in this way. A score of less than 30 mm is considered mild pain, between 31 and 54 mm, moderate, and 55 mm, severe.

SECONDARY OUTCOMES:
Change in Pain Severity | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  To assess the severity of pain, it will be used. the Spanish version of the chronic pain grading scale (EGDC), which is divided into two subscales (the first evaluates the intensity of pain and the second the disability perceived with the first subscale). The Spanish version has proven to be valid and reliable for assessing the severity of chronic pain. The total score that can be obtained ranges from 0 to 70 points, and can generate 5 graduation levels, from less serious to more serious
Change in Neck Disability | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  Validated version in Spanish of the "Neck Disability Index". It measures the level of disability perceived by the patient as a consequence of their neck pain. It consists of 10 elements, related to functional activities of daily living, pain intensity, concentration capacity, work capacity and headache. . The total score ranges from 0 (good function) to 50 (disability). In general, a score between 5 and 14 is considered a mild disability, between 15 and 24 moderate disabilities and 25 severe disabilities.
Change in Strait State Anxiety | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  We will use the version adapted to Spanish of the State Scale (STAI-E) of the "State-Trait Anxiety Inventory" (STAI). The total scores for each of the subscales range between 0 and 60 points. Specifically, STAI-E is suitable for assessing state anxiety in a wide variety of clinical situations. In addition, it has good reliability and previously demonstrated validity.
Chage in Pain Related Anxiety | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  abbreviated version of the PASS scale ("The Pain Anxiety Symptoms Scale"). It consists of 20 items that measure 4 anxiety components before pain: fear, escape/avoidance, cognitive anxiety, and physiological anxiety. Patients rate each of the items using a 6-point Likert scale; be 0 never and 5 always. The total score ranges from 0 to 100.
Change in Catastrophizing | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  Spanish version of the "Catastrophizing Pain Scale" (PCS). It consists of 13 elements that eval.an catastrophic cognitive-emotional processes with respect to pain and collect the three main dimensions of catastrophism - rumination, increase (exaggeration of the unpleasantness of pain and pain). They are evaluated on a Likert scale. The total score range is between 0 and 52. The Spanish version of the PCS has shown good internal consistency
Change in Kinesiophobia | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  TAMPA SCALE OF KINESIOPHOBIA, TSK-11: allows to know the degree of fear of movement or re-injury. The validated Spanish version of the 11-position scale has a total score of 11 to 44 points and has two subscales: activity avoidance and harm. This scale has been shown to have good validity and reliability
Change in Fear of Pain | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  Questionnaire, FPQ-III: The purpose is to evaluate the emotional components of pain, the fears and apprehensions of an individual in the face of a varied nature of stimuli and situations that can cause pain. It will be used. The short version FPQ-SF (Short Form) of 9 points. The total score of the questionnaire fluctuate. between 30 and 150 points
Change in Depression | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  BECK DEPRESSION INVENTORY-II (BDI-II) It is the most widely used questionnaire worldwide and nationally to assess depression. We used the Spanish adaptation of the Beck II Depression Inventory. The total score ranges from 0 to 63 points. Regarding the cut-off point, a specific one cannot be established, since it depends on the population studied and the purpose of the study, but it ranges between 12 and 19 to indicate the presence of depressive symptoms. It has been seen that a change of 5 points in the Beck Depression Inventory can be a reasonable estimate of a CID
Change in Quality of Life | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The quality of life of patients is measured. with the EuroQoL-5D questionnaire (EQ-5D), 5 factors: mobility, personal care, daily activities, pain/discomfort and anxiety/depression, with a theoretical range of 1 to 5 in each factor that responds to five levels of severity, in which higher scores represent more serious health conditions. A second element consisting of a vertical VAS with a theoretical range from 0 (the worst imaginable health state) to 100 points (the best imaginable health state). The EQ-5D has presented good psychometric characteristics
Change in Fatigue after deep neck flexors Test | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The deep neck flexor strength test (DNFR) and the fatigue visual analog scale (FVAS) were used. to measure the resistance and the subjective sensation of fatigue in the deep flexors of the neck.
Change in Cervical Range of Motion | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  It will be evaluated using the CROM (Cervical Range of Motion) device. It consists of 3 inclinometers attached to a lightweight plastic frame, secured with Velcro straps for closure. The protocol used will be A sequence of 3 measurements, with an interval of 30 seconds between each measurement
Change in Pain Pressure Treshold | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  A digital algometer (FDX 25, Wagner Instruments, Greenwich, CT, USA) will be used, consisting of a rubber head (1 cm2), attached to a manometer
Change in Conditioned Pain Modulation | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  We will perform the provocation of accessory pain through the tourniquet test with a pneumatic cuff placed on the arm, inflated until the first sensation of pain, waiting 30 seconds, and the subject is asked to evaluate the level of subjective pain. in a GO
Change in Central Sensitization | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  CENTRAL SENSITIZATION INVENTORY (CSI): Used to identify symptoms related to central sensitization. Formed by 25 elements (maximum of 100). The results are interpreted: subclinical from 0 to 29; mild from 30 to 39; moderate from 40 to 49; severe from 50 to 59; and extreme from 60 to 100. The Spanish version will be used

OTHER OUTCOMES:
Patient Satisfaction | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The Global Assessment of Change (GROC) is the questionnaire that we will use to find out the patients' satisfaction with the general results of the treatments used in our study. The GROC is a 15-point scale whose central value is 0 (no change), above or to the left we find values that go from -1 to -7 (much worse) and below or to the right from +1 to + 7 (much worse). better)
Drug Consumption | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The type and average consumption of drugs per week will be recorded. at the baseline visit (consumption in the month before starting the intervention) and at the follow-up visits.
Days of Sick Leave | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  All days that patients have not been to work and are unable to go to work will be counted to calculate sick leave days.
Adherence to treatment | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  It will register. patient attendance at treatment sessions. Attending 3 of the 5 sessions is considered adequate adherence. Adhesion will be calculated. as the ratio of the number of treatment sessions that were carried out in relation to the number of sessions prescribed.
Assessment of adverse effects | Up to 1 week before the intervention, up to 1 day after the intervention, and at 3, 6 and 12 months after intervention
  The participants will be asked about all the possible adverse effects, they will be recorded in a questionnaire that will be collected from the patients after receiving the different treatments, and serious adverse effects will be reported to the research committee of the health care centers.
Therapeutic Alliance in Physiotherapy | After half of the treatment and after the treatment
  The spanish version of the therapeutic alliance in physiotherapy questionnaire will be used (CAF-P). It is a 14 item scale in which each is assessed on a three item likert like scale from totally disagree ( 2 points), partially disagree (1 point), neither agree or disagree (0 points), partially agree (3 points), and totally agree (4 points). Reaching a maximun of 56 points which means excellent therapeutic alliance and 0 point being the minimun, meaning no alliance.

CONTACTS AND LOCATIONS:
Overall Officials: María Adoración Prieto Aldana, 1st, Principal Investigator — Gerencia de Atención Primaria de la Comunidad de Madrid
Locations (1):
- Gerencia de Atención Primaria de la Comunidad de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Due to the data protection law the information about individuals will be kept under a password in an electronic data protection website. After 2 years it may be made available under request.

REFERENCES:
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S39-51. doi: 10.1097/BRS.0b013e31816454c8. PMID 18204398
- [Background] Palacios-Cena D, Alonso-Blanco C, Hernandez-Barrera V, Carrasco-Garrido P, Jimenez-Garcia R, Fernandez-de-las-Penas C. Prevalence of neck and low back pain in community-dwelling adults in Spain: an updated population-based national study (2009/10-2011/12). Eur Spine J. 2015 Mar;24(3):482-92. doi: 10.1007/s00586-014-3567-5. Epub 2014 Sep 11. PMID 25208501
- [Background] Hoving JL, Koes BW, de Vet HC, van der Windt DA, Assendelft WJ, van Mameren H, Deville WL, Pool JJ, Scholten RJ, Bouter LM. Manual therapy, physical therapy, or continued care by a general practitioner for patients with neck pain. A randomized, controlled trial. Ann Intern Med. 2002 May 21;136(10):713-22. doi: 10.7326/0003-4819-136-10-200205210-00006. PMID 12020139
- [Background] Bogduk N. The anatomy and pathophysiology of neck pain. Phys Med Rehabil Clin N Am. 2011 Aug;22(3):367-82, vii. doi: 10.1016/j.pmr.2011.03.008. PMID 21824580
- [Background] Gerrits MMJG, van Oppen P, van Marwijk HWJ, Penninx BWJH, van der Horst HE. Pain and the onset of depressive and anxiety disorders. Pain. 2014 Jan;155(1):53-59. doi: 10.1016/j.pain.2013.09.005. Epub 2013 Sep 6. PMID 24012953
- [Background] Borghouts JAJ, Koes BW, Vondeling H, Bouter LM. Cost-of-illness of neck pain in The Netherlands in 1996. Pain. 1999 Apr;80(3):629-636. doi: 10.1016/S0304-3959(98)00268-1. PMID 10342424
- [Background] D'Sylva J, Miller J, Gross A, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; Cervical Overview Group. Manual therapy with or without physical medicine modalities for neck pain: a systematic review. Man Ther. 2010 Oct;15(5):415-33. doi: 10.1016/j.math.2010.04.003. Epub 2010 Jun 9. PMID 20538501
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644
- [Background] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Background] Sterling M, Jull G, Wright A. Cervical mobilisation: concurrent effects on pain, sympathetic nervous system activity and motor activity. Man Ther. 2001 May;6(2):72-81. doi: 10.1054/math.2000.0378. PMID 11414776
- [Background] Fernandez-de-las-Penas C, Palomeque-del-Cerro L, Rodriguez-Blanco C, Gomez-Conesa A, Miangolarra-Page JC. Changes in neck pain and active range of motion after a single thoracic spine manipulation in subjects presenting with mechanical neck pain: a case series. J Manipulative Physiol Ther. 2007 May;30(4):312-20. doi: 10.1016/j.jmpt.2007.03.007. PMID 17509440
- [Background] O'Leary S, Falla D, Hodges PW, Jull G, Vicenzino B. Specific therapeutic exercise of the neck induces immediate local hypoalgesia. J Pain. 2007 Nov;8(11):832-9. doi: 10.1016/j.jpain.2007.05.014. Epub 2007 Jul 19. PMID 17644487
- [Background] Oostendorp RA, Elvers H, Mikolajewska E, Laekeman M, van Trijffel E, Samwel H, Duquet W. Manual physical therapists' use of biopsychosocial history taking in the management of patients with back or neck pain in clinical practice. ScientificWorldJournal. 2015;2015:170463. doi: 10.1155/2015/170463. Epub 2015 Apr 5. PMID 25945358
- [Background] Crossley KM, Vicenzino B, Lentzos J, Schache AG, Pandy MG, Ozturk H, Hinman RS. Exercise, education, manual-therapy and taping compared to education for patellofemoral osteoarthritis: a blinded, randomised clinical trial. Osteoarthritis Cartilage. 2015 Sep;23(9):1457-64. doi: 10.1016/j.joca.2015.04.024. Epub 2015 May 7. PMID 25960116
- [Background] Tellez-Garcia M, de-la-Llave-Rincon AI, Salom-Moreno J, Palacios-Cena M, Ortega-Santiago R, Fernandez-de-Las-Penas C. Neuroscience education in addition to trigger point dry needling for the management of patients with mechanical chronic low back pain: A preliminary clinical trial. J Bodyw Mov Ther. 2015 Jul;19(3):464-72. doi: 10.1016/j.jbmt.2014.11.012. Epub 2014 Nov 22. PMID 26118519
- [Background] Meeus M, Nijs J, Hamers V, Ickmans K, Oosterwijck JV. The efficacy of patient education in whiplash associated disorders: a systematic review. Pain Physician. 2012 Sep-Oct;15(5):351-61. PMID 22996847
- [Background] Gross A, Forget M, St George K, Fraser MM, Graham N, Perry L, Burnie SJ, Goldsmith CH, Haines T, Brunarski D. Patient education for neck pain. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD005106. doi: 10.1002/14651858.CD005106.pub4. PMID 22419306
- [Background] Haines T, Gross AR, Burnie S, Goldsmith CH, Perry L, Graham N; Cervical Overview Group (COG). A Cochrane review of patient education for neck pain. Spine J. 2009 Oct;9(10):859-71. doi: 10.1016/j.spinee.2009.04.019. Epub 2009 Jul 12. PMID 19596214
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Meeus M, Nijs J, Van Oosterwijck J, Van Alsenoy V, Truijen S. Pain physiology education improves pain beliefs in patients with chronic fatigue syndrome compared with pacing and self-management education: a double-blind randomized controlled trial. Arch Phys Med Rehabil. 2010 Aug;91(8):1153-9. doi: 10.1016/j.apmr.2010.04.020. PMID 20684894
- [Background] Louw A, Butler DS, Diener I, Puentedura EJ. Development of a preoperative neuroscience educational program for patients with lumbar radiculopathy. Am J Phys Med Rehabil. 2013 May;92(5):446-52. doi: 10.1097/PHM.0b013e3182876aa4. PMID 23478459
- [Background] Nijs J, Roussel N, Paul van Wilgen C, Koke A, Smeets R. Thinking beyond muscles and joints: therapists' and patients' attitudes and beliefs regarding chronic musculoskeletal pain are key to applying effective treatment. Man Ther. 2013 Apr;18(2):96-102. doi: 10.1016/j.math.2012.11.001. Epub 2012 Dec 28. PMID 23273516
- [Background] Louw A, Diener I, Landers MR, Puentedura EJ. Preoperative pain neuroscience education for lumbar radiculopathy: a multicenter randomized controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2014 Aug 15;39(18):1449-57. doi: 10.1097/BRS.0000000000000444. PMID 24875964
- [Background] Nijs J, Wijma AJ, Willaert W, Huysmans E, Mintken P, Smeets R, Goossens M, van Wilgen CP, Van Bogaert W, Louw A, Cleland J, Donaldson M. Integrating Motivational Interviewing in Pain Neuroscience Education for People With Chronic Pain: A Practical Guide for Clinicians. Phys Ther. 2020 May 18;100(5):846-859. doi: 10.1093/ptj/pzaa021. PMID 31995191
- [Derived] Morales Tejera D, Nijs J, Malfliet A, Prieto Aldana MA, Gallardo Vidal MI, Polentinos Castro E, Linares Fernandez MT, Fernandez-Carnero J. Effectiveness of pain neuroscience education, motivational interviewing and cognition targeted exercise therapy in patients with chronic neck pain: protocol for a multicentre randomised controlled trial (the COGMO-AP study). BMJ Open. 2025 Feb 20;15(2):e087788. doi: 10.1136/bmjopen-2024-087788. PMID 39979041